CLINICAL TRIAL: NCT00110916
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Intra-Articular metHuIL-1ra (Anakinra) in Subjects With Osteoarthritis (OA) of the Knee
Brief Title: Treatment for Patients With Osteoarthritis (OA) of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20040100
Record Dates: First submitted 2005-05-16; First posted 2005-05-17 (Estimated); Last update posted 2008-02-22 (Estimated); Status verified 2008-02

CONDITIONS: Osteoarthritis
Keywords: Intra-articular; Osteoarthritis; OA; anakinra; Amgen
MeSH Terms: conditions — Osteoarthritis | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Anakinra (Experimental): anakinra
  Interventions: Drug: Intra-articular metHuIL-1ra (anakinra)
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Intra-articular metHuIL-1ra (anakinra) — anakinra
  Arms: Anakinra
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the clinical response in subjects with symptomatic OA of the knee following a single 50 mg anakinra, 150 mg anakinra or placebo intra-articular (IA) injection.

ELIGIBILITY:
Inclusion Criteria: - Diagnosed with knee OA as determined by American College of Rheumatology (ACR) criteria - Pain defined by a level of greater than 30 mm on a 100 mm Visual Analogue Scale (VAS) - No evidence of active effusion or inflammatory flare, confirmed by investigator - Must exhibit radiographic evidence of tibio-femoral compartment knee OA within 12 months of screening - Stable doses of any non-prescribed supplements (e.g. glucosamine or chondroitin sulphate, shark cartilage, diacerhein, soya extract) for at least 2 months prior to screening - Unchanged use of physical therapy, biomechanical devices or orthotic support within at least 2 months of screening - Subjects on nonsteroidal anti-inflammatory drug (NSAID) therapy must discontinue NSAIDs 3 days prior to baseline (Day 1) - Before any study-specific procedure is performed, the appropriate written informed consent for participation in the study must be obtained Exclusion Criteria: - Malignancy within the previous 5 years, except for basal cell or in situ cancer - Significant hematologic disease - Active infection or history of recurrent or chronic infections - Known diagnosis of HIV, hepatitis B, or hepatitis C infection - Uncontrolled diabetes or cardiovascular disease and hypertension - Inflammatory arthropathy including secondary OA - Isolated OA of the patellofemoral joint (bi or tri-compartmental involvement are not exclusions) - End-stage ("bone-on-bone") OA (Kellgren Lawrence score of 4) - OA of the hip ipsilateral to the index knee - Total white cell count less than 2.0 x 109/L and/or platelet count less than 100 x 109/L observed within 1 month preceding screening - Prior IA injection of anakinra or experimental interleukin-1 (IL-1) inhibitor therapy - Concurrent treatment with subcutaneous (SC) anakinra - Concurrent or recent (less than or equal to 1 month) use of experimental therapy - Prior IA corticosteroid injection within 1 month of study - Prior viscosupplement therapy within 3 months of study - Contraindication(s) to IA injections - Subjects who are pregnant or breast-feeding, or plan to become pregnant during the study - Subject is not using adequate contraception - Known allergy to E coli-derived products - Unable to understand informed consent - Concerns regarding subject's compliance with the protocol procedures - Subject will not be available for follow-up assessment - Active substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2004-06; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
WOMAC | 12 weeks

SECONDARY OUTCOMES:
Pain Patient's global assessment | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Chevalier X, Goupille P, Beaulieu AD, Burch FX, Bensen WG, Conrozier T, Loeuille D, Kivitz AJ, Silver D, Appleton BE. Intraarticular injection of anakinra in osteoarthritis of the knee: a multicenter, randomized, double-blind, placebo-controlled study. Arthritis Rheum. 2009 Mar 15;61(3):344-52. doi: 10.1002/art.24096. PMID 19248129
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/20040100.pdf